CLINICAL TRIAL: NCT00002314
Title: A Phase II Study of Oral Ro 24-7429 (Tat Antagonist) in Patients With HIV-Related Kaposi's Sarcoma
Brief Title: A Study of Ro 24-7429 in Patients With HIV-Related Kaposi's Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 128A
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1993-12

CONDITIONS: Sarcoma, Kaposi; HIV Infections
Keywords: Sarcoma, Kaposi; Acquired Immunodeficiency Syndrome; Antineoplastic Agents; Gene Products, tat
MeSH Terms: conditions — Sarcoma, Kaposi; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Ro 24-7429

INTERVENTIONS:
Drug: Ro 24-7429

SUMMARY:
To study the effects of Ro 24-7429 on tumor growth in patients with HIV-related Kaposi's sarcoma. To study the safety and tolerance, effects on HIV replication, and immunologic effects of Ro 24-7429 in this patient population. To explore relationships between exposure to Ro 24-7429 and its metabolites with its antitumor and antiviral activities and drug toxicity.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV seropositivity.
* Biopsy-proven mucocutaneous Kaposi's sarcoma with fewer than 50 skin lesions and measurable disease.
* No active opportunistic infection. NOTE:
* Patients with CD4 count >= 200 cells/mm3 must have no prior opportunistic infection, as well as no active opportunistic infection.
* Life expectancy of at least 24 weeks.
* Stable weight (+/- 2 kg) by 28 days prior to study entry.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Other active malignancies (except basal cell carcinoma of the skin and in situ cervical cancer).
* Known or suspected hypersensitivity to benzodiazepines.
* Evidence of clinically significant cardiac, respiratory, hepatic, gastrointestinal, endocrine, hematologic, psychiatric, neurologic, dermatologic, or allergic disease as determined by the investigator.
* Ongoing diarrhea (> two liquid stools per day).
* Grade 2 or worse signs and symptoms of AIDS Dementia Complex.
* Alteration of mental status that may interfere with study compliance.

Concurrent Medication:

Excluded:

* AZT, ddI, or ddC.
* Experimental antiretrovirals.
* Biologic response modifiers or immunomodulating agents (e.g., interferon).
* Colony stimulating factors (erythropoietin, GM-CSF, G-CSF).
* Ganciclovir.
* Foscarnet.
* H-2 antagonists (cimetidine, ranitidine, famotidine, nizatidine).
* Omeprazole.
* Benzodiazepines.
* Any other investigational compound.
* Ongoing systemic treatment with corticosteroids (other than replacement therapy for adrenal insufficiency or short-term therapy of no more than 28 days for bronchial asthma).
* Cytotoxic chemotherapy (systemic and local).
* Drugs known to cause systemic toxicity, if avoidable (e.g., myelosuppressive, hepatotoxic, nephrotoxic, or neurotoxic drugs).
* Paromomycin sulfate.
* Chronic suppressive therapy for CMV and/or MAI.

Patients with the following prior condition are excluded:

History of serious adverse reactions to benzodiazepines.

Prior Medication:

Excluded:

* Interferons or immune modulators within 4 weeks prior to study entry.
* Prior systemic cytotoxic chemotherapy (patients with CD4 counts >= 200 cells/mm3 only).
* Benzodiazepines within 14 days prior to study entry.
* Intralesional chemotherapy for Kaposi's sarcoma within 2 weeks prior to study entry.
* Therapy with antiretroviral drugs (including AZT, ddI, ddC, d4T) or investigational drugs within 14 days prior to study entry.

Localized radiotherapy. Radiotherapy (other than localized). Active drug or alcohol abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - CARE Ctr / UCLA Med Ctr, Los Angeles, California
  - New England Deaconess Hosp, Boston, Massachusetts